CLINICAL TRIAL: NCT03540862
Title: Negative Pressure Ventilator in Long-term Pulmonary Rehabilitation for Chronic Obstructive Pulmonary Disease: Outcome Analysis
Brief Title: Negative Pressure Ventilator in Long-term Pulmonary Rehabilitation for Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201600035A3
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic obstructive pulmonary disease; Maintenance Negative Pressure Ventilation- assisted pulmonary rehabilitation; Six minute walk test; Overall survival
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- NPV: a hospital-based maintenance NPV program including NPV support, breathing training and an educational program (relaxation techniques, and home pacing walking exercise) in daily clinical practice. Patients received NPV with breathing training via the cuirass ventilator (Philips Respironics Lifecare NEV-100) settings for 60 min. The ventilator was set to control model with frequency of 12 cycles/min, 30% of the ratio of inspiratory time to total breathing cycle time (Ti/Ttot) and delivered negative pressures ranging -20 to -30 cm H2O. In the NPV group, patients underwent the hospital-based NPV once every week as the maintenance program.
  Interventions: Device: maintenance negative pressure ventilation (Philips Respironics Lifecare NEV-100)
- Control: If patients do not wish to enter the hospital-based NPV program, they are placed in the control group and are trained to perform breathing training, relaxation techniques and home pacing walking exercise.

INTERVENTIONS:
Device: maintenance negative pressure ventilation (Philips Respironics Lifecare NEV-100) — hospital-based NPV once every week as the maintenance program
  Groups: NPV

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by irreversible airflow obstruction with chronic airway inflammation and emphysematous changes in the lung parenchyma, thus leading to air-trapping, as well as extional dyspnea. The investigators have previously observed that NPV used as an adjuvant to pulmonary rehabilitation improves lung function, exercise capacity, and reduces exacerbations. The investigators now sought to determine whether long-term maintenance NPV improves long-term clinical outcomes and reduces mortality in COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by irreversible airflow obstruction with chronic airway inflammation and emphysematous changes in the lung parenchyma, thus leading to air-trapping, as well as extional dyspnea. The mechanism underlying desaturation during 6MWT in patients with COPD is multifactorial involving dynamic hyperinflation and impaired gas exchange that worsens ventilation-perfusion mismatch. Previous studies have shown that oxygen desaturation during the 6MWT predicts mortality and increases the risk of adverse outcomes in COPD patients. However, there is a paucity of studies that have looked at effective treatments to counter the consequences of hypoxemia during exertion.

The investigators have established a hospital-based maintenance pulmonary rehabilitation program together with NPV for COPD, and the investigators have shown that the benefits of NPV improves lung function and exercise capacity, and reduces acute exacerbation and medical costs. The investigators now sought to determine whether long-term maintenance NPV improves long-term clinical outcomes and reduces mortality in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Main diagnosis of Chronic Obstructive Pulmonary Disease
* Stable status at enrollment
* Able to come to pulmonary rehab center

Exclusion Criteria:

* Infection or acute excerbation condition at enrollment
* Severe neuromuscular, cardiac disease or dementia
* Unable to perform six minute walk test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from the outpatient clinic of Chang Gung Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2003-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall mortality | 8 years
  Death of all causes
COPD-related mortality | 8 years
  pulmonary, lung cancer and cardiovascular death

SECONDARY OUTCOMES:
Lung function | 8 years
  forced expiratory volume in one second (FEV1)
6 minute walking distance | 8 years
  6 minute walking test distance
Severe exacerbations | 8 years
  ER visits or hospitalisations

CONTACTS AND LOCATIONS:
Overall Officials: Hung yu Huang, MD, Principal Investigator — chang gung hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan (r.o.c.), Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang HY, Chou PC, Joa WC, Chen LF, Sheng TF, Lin HC, Yang LY, Pan YB, Chung FT, Wang CH, Kuo HP. Pulmonary rehabilitation coupled with negative pressure ventilation decreases decline in lung function, hospitalizations, and medical cost in COPD: A 5-year study. Medicine (Baltimore). 2016 Oct;95(41):e5119. doi: 10.1097/MD.0000000000005119. PMID 27741132
- [Result] Gorini M, Corrado A, Villella G, Ginanni R, Augustynen A, Tozzi D. Physiologic effects of negative pressure ventilation in acute exacerbation of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Jun;163(7):1614-8. doi: 10.1164/ajrccm.163.7.2012079. PMID 11401883
- [Result] Waatevik M, Johannessen A, Gomez Real F, Aanerud M, Hardie JA, Bakke PS, Lind Eagan TM. Oxygen desaturation in 6-min walk test is a risk factor for adverse outcomes in COPD. Eur Respir J. 2016 Jul;48(1):82-91. doi: 10.1183/13993003.00975-2015. Epub 2016 Apr 13. PMID 27076586